CLINICAL TRIAL: NCT05559905
Title: A Phase 2a Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of MK-4482 in Healthy Participants Inoculated With Experimental Respiratory Syncytial Virus
Brief Title: Respiratory Syncytial Virus (RSV) Human Challenge Study of Molnupiravir in Healthy Participants (MK-4482-017)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4482-017; MK-4482-017 (Other: Merck)
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Syncytial Virus
MeSH Terms: interventions — molnupiravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Panel A: Molnupiravir Prophylaxis (Experimental): Participants received molnupiravir 800 mg every 12 hours for 5 days beginning on Day -1, and are inoculated with RSV-A Memphis 37b on Day 0. Participants switch to placebo beginning on the evening of Day 4 to the morning of Day 10.
  Interventions: Drug: Molnupiravir; Drug: Placebo; Biological: RSV A Memphis 37b
- Panel B: Molnupiravir Triggered Treatment (Experimental): Participants received placebo on Day -1, are inoculated with RSV-A Memphis 37b on Day 0, and continue to receive placebo until testing positive for RSV. Participants then received 800 mg of molnupiravir every 12 hours for 5 days.
  Interventions: Drug: Molnupiravir; Drug: Placebo; Biological: RSV A Memphis 37b
- Panel C: Matched Placebo (Placebo Comparator): Participants received placebo beginning on Day -1, are inoculated with RSV-A Memphis 37b on Day 0, and continue receiving placebo until the morning of Day 10.
  Interventions: Drug: Placebo; Biological: RSV A Memphis 37b

INTERVENTIONS:
Drug: Molnupiravir — Four molnupiravir 200 mg capsules (800 mg total dose) taken twice daily by mouth.
  Other Names: MK-4482
  Arms: Panel A: Molnupiravir Prophylaxis; Panel B: Molnupiravir Triggered Treatment
Drug: Placebo — Placebo capsule matched to molnupiravir taken twice daily by mouth.
Biological: RSV A Memphis 37b — RSV A Memphis 37b viral challenge given once by intranasal administration at a dosage of ~4 Log10 plaque forming units (PFUs).

SUMMARY:
This is a study of molnupiravir (MK-4482) in healthy participants who have been inoculated with an experimental Respiratory Syncytial Virus (RSV) [RSV-A Memphis 37b]. It is hypothesized that treatment with the drug MK-4482 (molnupiravir) will reduce the peak viral load (PVL) in the participant compared to placebo when given either before or after RSV-A Memphis 37b inoculation.

DETAILED DESCRIPTION:
Participants arrive at the study center for check-in between Day -3 and Day -1. Participants receive the assigned treatment beginning on Day -1. On Day 0, all participants receive viral inoculation with RSV-A Memphis 37b. All participants depart on Day 12 and follow-up is continued until Day 28.

The study is designed with the following arms:

* Panel A: Molupiravir Prophylaxis - in this arm, participants receive molupiravir beginning on Day -1, are incoluated with RSV-A Memphis 37b on Day 0, and continue receiving molnupiravir for a total of 5 days before switching to placebo through Day 10.
* Panel B: Molupiravir Triggered Treatment - in this arm, participants receive placebo beginning on Day -1 until testing positive for RSV. Participants are inoculated with RSV-A Memphis 37b on Day 0. When participants test positive for RSV, they switch to molnupiravir for a total of 5 consecutive days before switching back to placebo through Day 10. If participants in this arm do not test positive for RSV by Day 5, they automatically switch to molnupiravir through Day 10.
* Panel C: Placebo - in this arm, all participants receive placebo beginning on Day -1, are inoculated with RSV-A Memphis 37b on Day 0, and continue receiving placebo through Day 10.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health based on medical history, physical examination, vital sign measurements, spirometry, and electrocardiograms (ECGs) performed before randomization.
* Has a total body weight ≥50 kg and Body Mass Index (BMI) ≥18 kg/m^2 and ≤35 kg/m^2.
* For males, agrees to abstain from heterosexual intercourse OR use contraception unless confirmed to be azoospermic during the study and for 90 days after.
* For females, is not pregnant or breastfeeding, AND is either not a woman of childbearing potential (WOCBP) or is a WOCBP AND uses a highly effective contraceptive (low user dependency OR a user dependent hormonal method in combination with a barrier method), has a negative highly sensitive pregnancy test at screening, and has medical, menstrual, and recent sexual activity history reviewed by the investigator to decrease risk of early undetected pregnancy.

Exclusion Criteria:

* Has a history of, or currently active, symptoms or signs suggestive of upper or lower respiratory tract infection within 4 weeks prior to the first study visit.
* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Has a history of resolved depression and/or anxiety 1 or more years ago may be included at the discretion of the investigator.
* Has a history of cancer (malignancy).
* Has a history of rhinitis (including hay fever) which is clinically active or history of moderate to severe rhinitis, or history of seasonal allergic rhinitis likely to be active at the time of inclusion into the study and/or requiring regular nasal corticosteroids on an at least weekly basis, within 30 days of admission to quarantine.
* Has a history of atopic dermatitis/eczema which is clinically severe and/or requiring moderate to large amounts of daily dermal corticosteroids.
* If the reporting physician has diagnosed migraine can be included, provided there are no associated neurological symptoms such as hemiplegia or visual loss.
* If there is a physician diagnosed mild Irritable Bowel Syndrome not requiring regular treatment, can be included at the discretion of the investigator.
* Uses or anticipates use during study of herbal supplements within 7 days prior to Viral Challenge, any cytochrome P450 (CYP450)-inhibiting medications within 21 days prior to Viral Challenge, any over-the-counter medications (eg, ibuprofen) within 7 days prior to Viral Challenge, or any systemic anti-viral administration within 4 weeks of Viral Challenge/first dosing of study medication.
* Has evidence of receipt of vaccine within the 4 weeks prior to the planned date of viral challenge/first dosing with study medication (whichever occurs first).
* Intends to receive any vaccine before the last study visit.
* Has received any investigational drug within 3 months or 5 half-lives (whichever is greater) prior to the planned date of viral challenge/first dosing with study medication (whichever occurs first).
* Has received ≥3 investigational drugs in the past 12 months.
* Has had a prior inoculation with a virus from the same family as the challenge virus.
* Has smoked ≥10 pack years at any time (one pack of 20 cigarettes a day for 10 years).
* Has a recent history or presence of alcohol addiction, or excessive use of alcohol (weekly intake in excess of 28 units alcohol; 1 unit being a half glass of beer, a small glass of wine or a measure of spirits), or excessive consumption of xanthine-containing substances (eg, daily intake in excess of 5 cups of caffeinated drinks such as coffee, tea, cola).
* Has a lifetime history of anaphylaxis and/or a lifetime history of severe allergic reaction.
* Has any significant abnormality altering the anatomy of the nose in a substantial way or nasopharynx that may interfere with the aims of the study and, in particular, any of the nasal assessments or viral challenge.
* Has any clinically significant history of epistaxis (large nosebleeds) within the last 3 months of the first study visit and/or history of being hospitalized due to epistaxis on any previous occasion.
* Has had any nasal or sinus surgery within 3 months of the first study visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- hVIVO Services ( Site 0001), London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Cheng MH, Mann AJ, Maas BM, Zhao T, Bevan M, Schaeffer AK, Liao LE, Catchpole AP, Hilbert DW, Aubrey Stoch S, De Anda CS. A Phase 2a, Randomized, Placebo-Controlled Human Challenge Trial to Evaluate the Efficacy and Safety of Molnupiravir in Healthy Participants Inoculated with Respiratory Syncytial Virus. Pulm Ther. 2025 Jun;11(2):285-304. doi: 10.1007/s41030-025-00289-z. Epub 2025 Apr 2. PMID 40175624
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the lower quartile for immunogenicity to the RSV A Memphis 37b as determined by a serum microneutralization assay were screened for eligibility for this study.
Groups:
- Panel A: Molnupiravir Prophylaxis: Participants received molnupiravir 800 mg every 12 hours for 5 days beginning on Day -1 and were inoculated with RSV-A Memphis 37b on Day 0. Participants switched to placebo beginning on the evening of Day 4 to the morning of Day 10.
- Panel B: Molnupiravir Triggered Treatment: Participants received placebo on Day -1, were inoculated with RSV-A Memphis 37b on Day 0, and continued to receive placebo until testing positive for RSV. Participants then received 800 mg of molnupiravir every 12 hours for 5 days.
- Panel C: Matched Placebo: Participants received placebo beginning on Day -1, were inoculated with RSV-A Memphis 37b on Day 0, and continued receiving placebo until the morning of Day 10.
Period: Overall Study
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Started | 40 | 36 | 40
Started Study Medication | 39 | 36 | 40
Completed | 38 | 36 | 40
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Not Reported | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo | Total
Number analyzed (Participants) | 40 | 36 | 40 | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.6 (5.4) | 28.7 (8.2) | 26.8 (6.9) | 27.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 17 | 45
  Male | 25 | 23 | 23 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 40 | 35 | 40 | 115
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 7 | 15
  White | 32 | 25 | 29 | 86
  More than one race | 1 | 4 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Panel A vs Panel C: Peak Viral Load (PVL) Determined by Viral Quantitative Culture
Description: PVL was defined as the maximum viral load during a specified time period. PVL determined by viral quantitative culture (plaque assay) was measured from Day 2 up to Day 12 (end of participant quarantine). PVL (on the log10 scale) of RSV A Memphis 37b determined by viral quantitative culture (plaque assay) between Day 2 and Day 12 am after intranasal inoculation (Day 0) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the model.
Time Frame: From Day 2 up to Day 12
Population: All randomized participants in Panel A or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, and had available PVL viral quantitative culture data. Per protocol, Panel B was not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 plaque forming units (PFU)/mL
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel C: Matched Placebo
Number analyzed (Participants) | 32 | 34
log10 plaque forming units (PFU)/mL | 2.55 [1.81 to 3.30] | 2.84 [2.12 to 3.57]
Statistical Analysis 1: Comparison: Panel A: Molnupiravir Prophylaxis vs Panel C: Matched Placebo; Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the model. The mean PVL in each group and the differences in mean PVL between MK-4482 and placebo and the corresponding 2- sided 95% CI were computed based on the linear model; Test type: Superiority; p = 0.578, ANOVA; Difference in Least Squares Mean = -0.29, 90% CI 2-sided [-1.16 to 0.58]

2. Primary Outcome: Panel B vs. Panel C: Area Under the Viral Load-time Curve (VL-AUC) Determined by Viral Quantitative Culture
Description: VL-AUC between Day 2 and Day 12 after intranasal inoculation (Day 0) was computed for each participant, based on RSV viral load determined by viral quantitative culture (plaque assay) from nasal wash samples collected twice daily (morning and evening). In order to calculate the AUC, the actual time that the assessment was collected was used within the AUC calculation. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only Panel B (treatment) and Panel C (placebo) were included in the model. For both panels, only the participants with RSV infection were included.
Time Frame: From Day 2 up to Day 12
Population: All randomized participants in Panel B or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, were determined to be RSV infected, and had available VL-AUC viral quantitative culture data. Per protocol, Panel A was not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: day*log10 PFU/mL
Arm/Group | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 20 | 25
day*log10 PFU/mL | 7.02 [3.91 to 10.14] | 9.72 [6.93 to 12.50]
Statistical Analysis 1: Comparison: Panel B: Molnupiravir Triggered Treatment vs Panel C: Matched Placebo; Per protocol, only Panel B (treatment) and Panel C (placebo) were included in the model. For both panels, only the participants with RSV infection were included in the analysis. The mean VL-AUC in each group and the differences in mean VL-AUC between MK-4482 and placebo and the corresponding 2-sided 95% CI were computed based on the linear model; Test type: Superiority; p = 0.201, ANOVA; Difference in Least Squares Mean = -2.69, 90% CI 2-sided [-6.17 to -0.79]

3. Secondary Outcome: All Panels: Number of Participants Who Experienced ≥1 Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced an AE is reported.
Time Frame: From Day -1 up to Day 28
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 39 | 36 | 40
Participants | 13 | 15 | 13

4. Secondary Outcome: All Panels: Number of Participants Who Experienced ≥1 Serious AE (SAE)
Description: An SAE is any untoward medical occurrence that, at any dose, results in death; is life-threatening; requires hospitalization or prolongs existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly or birth defect; or is another important medical event such as invasive/malignant cancers or substance abuse/dependency. The number of participants who experienced an SAE is reported.
Time Frame: From Day -1 up to Day 28
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 39 | 36 | 40
Participants | 0 | 0 | 0

5. Secondary Outcome: All Panels: Number of Participants Who Experienced ≥1 Viral Challenge-Related AE
Description: A viral challenge-related AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, that was considered related to the viral challenge (inoculation). The number of participants who experienced AEs related to the viral challenge from viral challenge (Day 0) up to the Day 28 follow-up is reported.
Time Frame: From Day 0 up to Day 28
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 39 | 36 | 40
Participants | 1 | 1 | 1

6. Secondary Outcome: All Panels: Number of Participants Who Experienced ≥1 Viral Challenge-Related SAE
Description: A viral challenge-related SAE was defined as any untoward medical occurrence that, at any dose, resulted in death; was life-threatening; required hospitalization or prolonged existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly or birth defect; or was another important medical event, that was considered related to the viral challenge (inoculation). The number of participants who experienced SAEs related to the viral challenge from viral challenge (Day 0) up to the Day 28 follow-up is reported.
Time Frame: From Day 0 up to Day 28
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 39 | 36 | 40
Participants | 0 | 0 | 0

7. Secondary Outcome: All Panels: Number of Participants Using Concomitant Medications From Viral Challenge Through Day 28
Description: Concomitant medications were defined as any prescription medications, over the counter drugs or dietary supplements that a participant happened to be taking while on study, in addition to molnupiravir. The number of participants using concomitant medications from viral challenge (Day 0) up through Day 28 is reported.
Time Frame: From Day 0 up to Day 28
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 39 | 36 | 40
Participants | 6 | 7 | 7

8. Secondary Outcome: Panel A vs. Panel C: VL-AUC Determined by Viral Quantitative Culture
Description: VL-AUC between Day 2 and Day 12 after intranasal inoculation (Day 0) was computed for each participant, based on RSV viral load determined by viral quantitative culture (plaque assay) from nasal wash samples collected twice daily (morning and evening). In order to calculate the AUC, the actual time that the assessment was collected was used within the AUC calculation. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the model.
Time Frame: From Day 2 up to Day 12
Population: All randomized participants in Panel A or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, and had available VL-AUC viral quantitative culture data. Per protocol, Panel B was not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: day*log10 PFU/mL
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel C: Matched Placebo
Number analyzed (Participants) | 32 | 34
day*log10 PFU/mL | 7.56 [4.95 to 10.17] | 8.17 [5.64 to 10.70]
Statistical Analysis 1: Comparison: Panel A: Molnupiravir Prophylaxis vs Panel C: Matched Placebo; Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the model. The mean VL-AUC in each group and the differences in mean VL-AUC between MK-4482 and placebo and the corresponding 2-sided 95% CI were computed based on the linear model; Test type: Superiority; p = 0.736, ANOVA; Difference in Least Squares Mean = -0.62, 90% CI 2-sided [-3.65 to 2.42]

9. Secondary Outcome: Panel A vs. Panel C: VL-AUC Determined by Real-time Quantitative Reverse Transcription Polymerase Chain Reaction (qRT-PCR)
Description: VL-AUC between Day 2 and Day 12 after intranasal inoculation (Day 0) was computed for each participant, based on RSV viral load determined by qRT-PCR from nasal wash samples collected twice daily (morning and evening). In order to calculate the AUC, the actual time that the assessment was collected was used within the AUC calculation. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the model.
Time Frame: Day 2 up through Day 12
Population: All randomized participants in Panel A or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into and who received the viral inoculation. Per protocol, Panel B was not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: day*log10 copies/mL
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel C: Matched Placebo
Number analyzed (Participants) | 38 | 39
day*log10 copies/mL | 17.62 [11.70 to 25.53] | 19.54 [13.70 to 25.39]
Statistical Analysis 1: Comparison: Panel A: Molnupiravir Prophylaxis vs Panel C: Matched Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.646, ANOVA; Difference in Least Squares Mean = -1.93, 90% CI 2-sided [-8.88 to 5.02]

10. Secondary Outcome: Panel A vs. Panel C: PVL Determined by qRT-PCR
Description: PVL was defined as the maximum viral load during a specified time period. PVL as determined by qRT-PCR was measured starting from Day 2 up to planned discharge from quarantine (Day 12 am). Nasal wash samples were collected and tested for RSV viral load by qRT-PCR twice daily from Day 2 through Day 11. A single nasal wash sample for RSV viral load by qRT-PCR was collected on Day 12. PVL by qRT-PCR was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the model.
Time Frame: Day 2 up through Day 12
Population: All randomized participants in Panel A or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, and had available PVL qRT-PCR data. Per protocol, Panel B was not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: day*log10 copies/mL
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel C: Matched Placebo
Number analyzed (Participants) | 38 | 39
day*log10 copies/mL | 4.66 [3.66 to 5.66] | 4.80 [3.81 to 5.79]
Statistical Analysis 1: Comparison: Panel A: Molnupiravir Prophylaxis vs Panel C: Matched Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.849, ANOVA; Difference in Least Squares Mean = -0.14, 90% CI 2-sided [-1.31 to 1.04]

11. Secondary Outcome: Panel A vs. Panel C: Area Under the Curve Over Time of Total Symptom Scores (TSS-AUC)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). Total symptom scores (TSS) ranged from 0 to 31, with higher scores indicating greater symptom severity. TSS were used to calculate the AUC for each participant based on the available non-missing calculated total symptom scores between Day -1 until Day 12 (quarantine discharge) using the Trapezoidal rule. TSS-AUC was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the model. TSS-AUC measured from 10 symptoms within the graded symptom scoring was reported.
Time Frame: From Day -1 up to Day 12
Population: All randomized participants in Panel A or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, and had available TSS data. Per protocol, Panel B was not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale*Days
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel C: Matched Placebo
Number analyzed (Participants) | 38 | 40
Scores on a Scale*Days | 7.5 [4.18 to 10.81] | 9.59 [6.36 to 12.82]
Statistical Analysis 1: Comparison: Panel A: Molnupiravir Prophylaxis vs Panel C: Matched Placebo; Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the model. The TSS-AUC in each group and the differences in mean TSS-AUC between MK-4482 and placebo and the corresponding 2- sided 95% CI were computed based on the linear model; Test type: Superiority; p = 0.371, ANOVA; Difference in Least Squares Mean = -2.09, 90% CI 2-sided [-5.97 to 1.78]

12. Secondary Outcome: Panel A vs. Panel C: Area Under the Curve Over Time of Total Symptom Scores Change From Baseline (TSS-AUC-CFB)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("absence") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. TSS were used to calculate the AUC for each participant based on the available non-missing calculated total symptom scores between Day -1 until Day 12 (quarantine discharge) using the Trapezoidal rule. TSS-AUC-CFB was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the model. TSS-AUC-CFB was defined as the change from baseline in TSS-AUC from Day -1 up to Day 12. TSS-AUC-CFB measured from 10 symptoms within the graded symptom scoring was reported.
Time Frame: Baseline (Day -1) and up to Day 12
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale*Days
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel C: Matched Placebo
Number analyzed (Participants) | 38 | 40
Scores on a Scale*Days | 6.84 [4.03 to 9.66] | 8.66 [5.92 to 11.41]
Statistical Analysis 1: Comparison: Panel A: Molnupiravir Prophylaxis vs Panel C: Matched Placebo; Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the model. The TSS-AUC-CFB in each group and the differences in mean TSS-AUC-CFB between MK-4482 and placebo and the corresponding 2- sided 95% CI were computed based on the linear model; Test type: Superiority; p = 0.360, ANOVA; Difference in Least Squares Mean = -1.82, 90% CI 2-sided [-5.11 to 1.47]

13. Secondary Outcome: Panel A vs. Panel C: Peak Total Symptom Scores
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. The highest TSS (defined as the sum of all 10 individual composite symptoms) was summarized by treatment group and analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the model. Peak TSS measured from 10 symptoms within the graded symptom scoring was reported.
Time Frame: From Day -1 up to Day 12
Population: as for outcome 11
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel C: Matched Placebo
Number analyzed (Participants) | 38 | 40
Scores on a Scale | 2.74 [1.85 to 3.62] | 3.20 [2.33 to 4.07]
Statistical Analysis 1: Comparison: Panel A: Molnupiravir Prophylaxis vs Panel C: Matched Placebo; Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the model. The mean peak TSS in each group and the differences in mean peak TSS between MK-4482 and placebo and the corresponding 2- sided 95% CI was computed based on the linear model; Test type: Superiority; p = 0.459, ANOVA; Difference in Least Squares Mean = -0.46, 90% CI 2-sided [-1.50 to 0.57]

14. Secondary Outcome: Panel A vs. Panel C: Peak Daily Symptom Score
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. The highest total symptom score recorded on each day, across the three assessments, for each participant was summarized descriptively by treatment group and assessment day. Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the analysis. Peak daily sums of symptom score measured from 10 symptoms within the graded symptom scoring were reported for Panels A and C.
Time Frame: From Day 2 up to Day 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel C: Matched Placebo
Number analyzed (Participants) | 38 | 40
Scores on a Scale
  Day 2 | 0.8 (1.13) | 1.1 (1.36)
  Day 3 | 0.6 (0.88) | 0.9 (1.24)
  Day 4 | 0.7 (0.98) | 1.0 (1.56)
  Day 5: number analyzed (Participants) | 38 | 39
  Day 5 | 0.8 (1.22) | 1.4 (1.90)
  Day 6: number analyzed (Participants) | 38 | 39
  Day 6 | 1.2 (1.41) | 2.1 (2.82)
  Day 7: number analyzed (Participants) | 38 | 39
  Day 7 | 1.4 (1.52) | 1.9 (3.02)
  Day 8: number analyzed (Participants) | 38 | 39
  Day 8 | 1.7 (2.24) | 1.8 (2.22)
  Day 9: number analyzed (Participants) | 38 | 39
  Day 9 | 1.4 (1.67) | 1.3 (1.90)
  Day 10: number analyzed (Participants) | 38 | 39
  Day 10 | 0.9 (1.83) | 0.8 (1.58)
  Day 11: number analyzed (Participants) | 38 | 39
  Day 11 | 0.7 (1.21) | 0.5 (1.02)
  Day 12: number analyzed (Participants) | 38 | 39
  Day 12 | 0.3 (0.76) | 0.3 (0.56)

15. Secondary Outcome: Panel A vs. Panel C: Percentage of Participants With Respiratory Syncytial Virus (RSV) Infection Based on qRT-PCR
Description: A qRT-PCR-confirmed RSV infection was defined as 2 quantifiable (≥ lower limit of quantification [LLOQ]) qRT-PCR measurements (reported on 2 or more independent samples over 2 days), from Day 2 up to Day 12. The number of participants with qRT-PCR-confirmed RSV infection is reported. Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the analysis.
Time Frame: From Day 2 up to Day 12
Population: All randomized participants in Panel A or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, and had available RSV infection qRT-PCR data. Per protocol, Panel B was not included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel C: Matched Placebo
Number analyzed (Participants) | 38 | 40
Percentage of Participants | 68.42 [51.35 to 82.50] | 65.00 [48.32 to 79.37]
Statistical Analysis 1: Comparison: Panel A: Molnupiravir Prophylaxis vs Panel C: Matched Placebo; Test type: Superiority; Difference in Percent (%) = 3.42, 95% CI 2-sided [-18.28 to 24.50]

16. Secondary Outcome: Panel A vs. Panel C: Percentage of Participants With RSV Infection Based on Cell Culture Measurement of Nasal Sample
Description: RSV infection based on cell culture measurement was defined as at least one positive (≥ LLOQ) cell culture measurement in nasal swab samples. The percentage of participants with at least one positive (≥ LLOQ) cell culture measurement in nasal swab samples is reported. Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the analysis.
Time Frame: From Day 2 up to Day 12
Population: All randomized participants in Panel A or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, and had at least 1 available positive RSV cell culture measurement data. Per protocol, Panel B was not included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel C: Matched Placebo
Number analyzed (Participants) | 38 | 40
Percentage of Participants | 57.89 [40.82 to 73.69] | 55.00 [38.49 to 70.74]
Statistical Analysis 1: Comparison: Panel A: Molnupiravir Prophylaxis vs Panel C: Matched Placebo; Test type: Superiority; Difference in Percent (%) = 2.89, 95% CI 2-sided [-19.37 to 25.69]

17. Secondary Outcome: Panel A vs. Panel C: Percentage of Participants With qRT-PCR Confirmed Symptomatic RSV Infection
Description: Symptomatic RSV infection was defined as 2 quantifiable (≥LLOQ) qRT-PCR measurements reported on 2 or more days and either one or more clinical symptoms of any grade from two different categories in the symptom scoring system (upper respiratory, lower respiratory, systemic) or one grade 2 symptom from any category. The percentage of participants with qRT-PCR-confirmed symptomatic RSV infection is reported. Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the analysis.
Time Frame: From Day 2 up to Day 12
Population: All randomized participants in Panel A or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, and had available RSV symptomatic infection data. Per protocol, Panel B was not included in this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel C: Matched Placebo
Number analyzed (Participants) | 38 | 40
Percentage of Participants | 47.37 [30.98 to 64.18] | 50.00 [33.80 to 66.20]
Statistical Analysis 1: Comparison: Panel A: Molnupiravir Prophylaxis vs Panel C: Matched Placebo; Test type: Superiority; Difference in Percent (%) = -2.63, 95% CI 2-sided [-25.07 to 19.91]

18. Secondary Outcome: Panel A vs. Panel C: Percentage of Participants With qRT-PCR Confirmed Moderately Severe Symptomatic RSV Infection
Description: Moderately severe symptomatic RSV infection was defined as 2 quantifiable (≥LLOQ) qRT-PCR measurements reported on 2 or more consecutive days and any symptom scores of grade ≥2 at a single time point. The percentage of participants with qRT-PCR-confirmed moderately severe symptomatic RSV infection is reported. Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the analysis.
Time Frame: From Day 2 up to Day 12
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel C: Matched Placebo
Number analyzed (Participants) | 38 | 40
Percentage of Participants | 26.32 [13.40 to 43.10] | 42.50 [27.04 to 59.11]
Statistical Analysis 1: Comparison: Panel A: Molnupiravir Prophylaxis vs Panel C: Matched Placebo; Test type: Superiority; Difference in Percent (%) = -16.18, 95% CI 2-sided [-36.77 to 5.64]

19. Secondary Outcome: Panel A vs. Panel C: Percentage of Participants With Culture-Confirmed Symptomatic RSV Infection
Description: Culture-confirmed symptomatic RSV infection was defined by 1 quantifiable (≥LLOQ) cell culture measurement from Day 2 up to Day 12, and either one or more clinical symptoms of any grade from two different categories in the symptom scoring system (upper respiratory, lower respiratory, systemic) or one grade 2 symptom from any category. The percentage of participants with culture confirmed symptomatic RSV infection is reported. Per protocol, only Panel A (prophylaxis) and Panel C (placebo) were included in the analysis.
Time Frame: From Day 2 up to Day 12
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel C: Matched Placebo
Number analyzed (Participants) | 38 | 40
Percentage of Participants | 42.11 [26.31 to 59.18] | 45.00 [29.26 to 61.51]
Statistical Analysis 1: Comparison: Panel A: Molnupiravir Prophylaxis vs Panel C: Matched Placebo; Test type: Superiority; Difference in Percent (%) = -2.89, 95% CI 2-sided [-25.69 to 19.37]

20. Secondary Outcome: Panel B vs. Panel C: PVL Determined by Viral Quantitative Culture
Description: PVL was defined as the maximum viral load during a specified time period. PVL as determined by viral quantitative culture was measured starting from Day 2 up to planned discharge from quarantine (Day 12 am). PVL (on the log10 scale) of RSV A Memphis 37b determined by viral quantitative culture (plaque assay) between Day 2 and Day 12 am after intranasal inoculation (Day 0) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only Panel B (treatment) and Panel C (placebo) are included in the model. For both panels, only the participants with RSV infection were included in the analysis.
Time Frame: From Day 2 up to Day 12
Population: All randomized participants in Panel B or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, were determined to be RSV infected, and had available PVL viral quantitative culture data. Per protocol, Panel A was not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 PFU/mL
Arm/Group | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 20 | 25
log10 PFU/mL | 2.85 [1.96 to 3.74] | 3.53 [2.74 to 4.33]
Statistical Analysis 1: Comparison: Panel B: Molnupiravir Triggered Treatment vs Panel C: Matched Placebo; Per protocol, only Panel B (treatment) and Panel C (placebo) are included in the model. For both panels, only the participants with RSV infection were included. The mean PVL in each group and the differences in mean PVL between MK-4482 and placebo and the corresponding 2- sided 95% CI were computed based on the linear model; Test type: Superiority; p = 0.253, ANOVA; Difference in Least Squares Mean = -0.69, 90% CI 2-sided [-1.68 to 0.31]

21. Secondary Outcome: Panel B vs. Panel C: Time to Negative Test by Viral Quantitative Culture
Description: The time to negative test was defined as length of time in days between the date and time of the first MK-4482 administration to the date and time of first confirmed negative test after peak viral culture measurement. A negative test is a result below the low limit of quantification (LLOQ) by viral quantitative culture (plaque assay). The Kaplan-Meier estimate median in days is reported. Per protocol, only Panel B (treatment) and Panel C (placebo) are included in the model. For both panels, only the participants with RSV infection were included in the analysis.
Time Frame: From Day 2 up to Day 12
Population: All randomized participants in Panel B or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, were determined to be RSV infected, and had available negative test by viral quantitative culture data. Per protocol, Panel A was not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 16 | 19
Days | 5.0 [4.0 to NA] — N/A: Upper limit of 95% confidence interval was not reached due to insufficient number of events (i.e. participants with negative test). | 5.0 [4.0 to 6.0]
Statistical Analysis 1: Comparison: Panel B: Molnupiravir Triggered Treatment vs Panel C: Matched Placebo; Test type: Superiority; p = 0.1708, Log Rank; Hazard Ratio (HR) = 1.72, 95% CI [0.83 to 3.57] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

22. Secondary Outcome: Panel B vs. Panel C: VL-AUC Determined by qRT-PCR
Description: VL-AUC between Day 2 and Day 12 after intranasal inoculation (Day 0) was computed for each participant, based on RSV viral load determined by qRT-PCR from nasal wash samples collected twice daily (morning and evening). In order to calculate the AUC, the actual time that the assessment was collected was used within the AUC calculation. VL-AUC (on the log10 scale) was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only Panel B (treatment) and Panel C (placebo) are included in the model. For both panels, only the participants with RSV infection were included in the analysis.
Time Frame: From Day 2 up to Day 12
Population: All randomized participants in Panel B or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, were determined to be RSV infected, and had available VL-AUC qRT-PCR data. Per protocol, Panel A was not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: days*log10 copies/mL
Arm/Group | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 23 | 26
days*log10 copies/mL | 20.58 [13.00 to 28.16] | 26.51 [19.38 to 33.64]
Statistical Analysis 1: Comparison: Panel B: Molnupiravir Triggered Treatment vs Panel C: Matched Placebo; Per protocol, only Panel B (treatment) and Panel C (placebo) are included in the model. For both panels, only the participants with RSV infection were included in the analysis. The mean VL-AUC in each group and the differences in mean VL-AUC between MK-4482 and placebo and the corresponding 2-sided 95% CI were computed based on the linear model; Test type: Superiority; p = 0.257, ANOVA; Difference in Least Squares Mean = -5.93, 90% CI 2-sided [-14.61 to 2.75]

23. Secondary Outcome: Panel B vs. Panel C: PVL Determined by qRT-PCR
Description: PVL was defined as the maximum viral load during a specified time period. PVL as determined by qRT-PCR was measured starting from Day 2 up to planned discharge from quarantine (Day 12 am). Nasal wash samples were collected and tested for RSV viral load by qRT-PCR twice daily from Day 2 through Day 11. A single nasal wash sample for RSV viral load by qRT-PCR was collected on Day 12. PVL by qRT-PCR were analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only Panel B (treatment) and Panel C (placebo) are included in the model. For both panels, only the participants with RSV infection were included in the analysis.
Time Frame: From Day 2 up to Day 12
Population: All randomized participants in Panel B or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, were determined to be RSV infected, and had available PVL qRT-PCR data. Per protocol, Panel A was not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 PFU/mL
Arm/Group | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 23 | 26
log10 PFU/mL | 5.43 [4.30 to 6.56] | 6.02 [4.95 to 7.08]
Statistical Analysis 1: Comparison: Panel B: Molnupiravir Triggered Treatment vs Panel C: Matched Placebo; Per protocol, only Panel B (treatment) and Panel C (placebo) are included in the model. For both panels, only the participants with RSV infection were included in the analysis. The mean PVL in each group and the differences in mean PVL between MK-4482 and placebo and the corresponding 2- sided 95% CI were computed based on the linear model; Test type: Superiority; p = 0.453, ANOVA; Difference in Least Squares Mean = -0.58, 90% CI 2-sided [-1.88 to 0.71]

24. Secondary Outcome: Panel B vs. Panel C: Time to Negative Test by qRT-PCR
Description: The time (days) to confirmed negative test by qRT-PCR was defined as the length of time between the date and time of the first investigational medicinal product (IMP) administration to the date and time of first confirmed undetectable (<LLOQ) qRT-PCR result after peak qRT-PCR measurement. The time to negative test starting at Day 2 to first confirmed undetectable (<LLOQ) assessment after peak measure is reported. Per protocol, only Panel B (treatment) and Panel C (placebo) are included in the model. For both panels, only the participants with RSV infection were included in the analysis.
Time Frame: From Day 2 up to Day 12
Population: All randomized participants in Panel B or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, were determined to be RSV infected, and had available negative test qRT-PCR data. Per protocol, Panel A was not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 20 | 24
Days | NA [6.0 to NA] — N/A: Upper limit of 95% confidence interval was not reached due to insufficient number of events (i.e. participants with negative test). | 9.0 [7.0 to NA] — N/A: Upper limit of 95% confidence interval was not reached due to insufficient number of events (i.e. participants with negative test).
Statistical Analysis 1: Comparison: Panel B: Molnupiravir Triggered Treatment vs Panel C: Matched Placebo; Test type: Superiority; p = 0.9121, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.44 to 2.51] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

25. Secondary Outcome: Panel B vs. Panel C: TSS-AUC
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). Total symptom scores (TSS) ranged from 0 to 31, with higher scores indicating greater symptom severity. TSS were used to calculate the AUC for each participant based on the available non-missing calculated total symptom scores between Day -1 until Day 12 (quarantine discharge) using the Trapezoidal rule. TSS-AUC was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only Panel B and Panel C are included in the model, and only participants with RSV infection were included in the analysis. TSS-AUC measured from 10 symptoms within the graded symptom scoring was reported.
Time Frame: From Day -1 up to Day 12
Population: All randomized participants in Panel B or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, were determined to be RSV infected, and had available TSS data. Per protocol, Panel A was not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale*Days
Arm/Group | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 23 | 26
Scores on a Scale*Days | 4.74 [1.76 to 7.72] | 6.57 [3.76 to 9.37]
Statistical Analysis 1: Comparison: Panel B: Molnupiravir Triggered Treatment vs Panel C: Matched Placebo; Per protocol, only Panel B (treatment) and Panel C (placebo) were included in the model. The TSS-AUC in each group and the differences in mean TSS-AUC between MK-4482 and placebo and the corresponding 2- sided 95% CI were computed based on the linear model; Test type: Superiority; p = 0.377, ANOVA; Difference in Least Squares Mean = -1.83, 90% CI 2-sided [-5.25 to 1.60]

26. Secondary Outcome: Panel B vs. Panel C: Area Under the Curve Over Time of Total Symptom Scores Change From Baseline (TSS-AUC-CFB)
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("absence") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. TSS were used to calculate the AUC for each participant based on the available non-missing calculated total symptom scores between Day -1 until Day 12 (quarantine discharge) using the Trapezoidal rule. TSS-AUC-CFB was analyzed using a linear model with treatment group as a fixed categorical effect. Per protocol, only Panel B and Panel C are included in the model, and only the participants with RSV infection were included in the analysis. TSS-AUC-CFB was defined as the change from baseline in TSS-AUC from Day -1 up to Day 12. TSS-AUC-CFB measured from 10 symptoms within the graded symptom scoring was reported.
Time Frame: Baseline (Day -1) and up to Day 12
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale*Days
Arm/Group | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 23 | 26
Scores on a Scale*Days | 2.60 [-1.02 to 6.23] | 2.74 [-0.67 to 6.15]
Statistical Analysis 1: Comparison: Panel B: Molnupiravir Triggered Treatment vs Panel C: Matched Placebo; Per protocol, only Panel B (treatment) and Panel C (placebo) were included in the model. The TSS-AUC-CFB in each group and the differences in mean TSS-AUC-CFB between MK-4482 and placebo and the corresponding 2- sided 95% CI were computed based on the linear model; Test type: Superiority; p = 0.958, ANOVA; Difference in Least Squares Mean = -0.13, 90% CI 2-sided [-4.28 to 4.02]

27. Secondary Outcome: Panel B vs. Panel C: Peak TSS
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. The highest total symptom score (defined as the sum of all 10 individual composite symptoms) was summarized by treatment group and analyzed using a linear model with treatment group as a fixed categorical effect. Peak TSS measured from 10 symptoms within the graded symptom scoring was reported for Panels B and C. Per protocol, only Panel B (treatment) and Panel C (placebo) are included in the model. For both panels, only the participants with RSV infection were included in the analysis.
Time Frame: From Day -1 up to Day 12
Population: as for outcome 25
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 23 | 26
Score on a Scale | 3.00 [1.61 to 4.39] | 3.62 [2.31 to 4.92]
Statistical Analysis 1: Comparison: Panel B: Molnupiravir Triggered Treatment vs Panel C: Matched Placebo; Per protocol, only Panel B (treatment) and Panel C (placebo) are included in the model. For both panels, only the participants with RSV infection were included in the analysis. The mean peak TSS in each group and the differences in mean peak TSS between MK-4482 and placebo and the corresponding 2- sided 95% CI was computed based on the linear model; Test type: Superiority; p = 0.520, ANOVA; Difference in Least Squares Mean = -0.62, 90% CI 2-sided [-2.21 to 0.98]

28. Secondary Outcome: Panel B vs. Panel C: Peak Daily Symptom Score
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. The highest total symptom score recorded on each day, across the three assessments, for each participant was summarized descriptively by treatment group and assessment day. Peak daily sums of symptom score measured from 10 symptoms within the graded symptom scoring were reported for Panels B and C. Per protocol, only Panel B (treatment) and Panel C (placebo) are included in the model. For both panels, only the participants with RSV infection were included in the analysis.
Time Frame: From Day -1 up to Day 12
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 23 | 26
Score on a Scale
  Day 1 | 0.6 (0.90) | 1.4 (1.6)
  Day 2 | 1.3 (1.89) | 2.0 (2.18)
  Day 3 | 1.5 (1.68) | 2.3 (2.31)
  Day 4 | 2.1 (2.44) | 2.7 (3.26)
  Day 5 | 1.8 (2.67) | 2.5 (3.37)
  Day 6 | 1.4 (2.29) | 1.5 (2.06)
  Day 7 | 0.7 (1.33) | 1.2 (2.12)
  Day 8 | 0.5 (1.08) | 0.7 (1.48)
  Day 9: number analyzed (Participants) | 6 | 13
  Day 9 | 1.0 (1.26) | 0.8 (1.42)
  Day 10: number analyzed (Participants) | 3 | 4
  Day 10 | 0.7 (1.15) | 0.5 (1.00)
  Day 11: number analyzed (Participants) | 2 | 1
  Day 11 | 1.0 (1.41) | 0.0 (0)

29. Secondary Outcome: Panel B vs. Panel C: Time to Symptom Resolution
Description: Participants used a symptom diary card to record the daily severity of 10 clinical symptoms on a scale ranging from 0 ("no symptoms") to 3 ("bothersome and interferes with activities"), with the exception of "shortness of breath" symptom which was scored from 0 ("no symptoms") to 4 ("symptoms at rest"). TSS ranged from 0 to 31, with higher scores indicating greater symptom severity. Symptom resolution was defined as a participant scoring 0 for the total symptom score for a 24-hour period (e.g., a minimum of three consecutive symptom diary cards, each with a score of 0 after their peak symptom score. The time in days to symptom resolution by treatment group, as measured from 10 symptoms within the graded daily symptom scoring system, was reported. Per protocol, only Panel B (treatment) and Panel C (placebo) are included in the model. For both panels, only the participants with RSV infection were included in the analysis.
Time Frame: From Day -1 up to Day 12
Population: All randomized participants in Panel B or Panel C who received 1 dose of the correct clinical material corresponding to the treatment group the participants were randomized into, who received the viral inoculation, were determined to be RSV infected, and had available symptom resolution data. Per protocol, Panel A was not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Days
Arm/Group | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
Number analyzed (Participants) | 17 | 18
Days | 6.0 [4.0 to 8.0] | 8.5 [6.0 to NA] — N/A: Upper limit of 95% confidence interval was not reached due to insufficient number of events (i.e. participants with negative test).
Statistical Analysis 1: Comparison: Panel B: Molnupiravir Triggered Treatment vs Panel C: Matched Placebo; Test type: Superiority; p = 0.0459, Log Rank; Two-sided p-value based on log-rank test; Hazard Ratio (HR) = 2.24, 95% CI 2-sided [0.99 to 5.07] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

30. Secondary Outcome: Panels A & B: Maximum Plasma Concentration (Cmax) of N-Hydroxycytidine (NHC)
Description: NHC is the pharmacologically active moiety of molnupiravir and therefore its primary pharmacokinetic measure. Cmax was defined as the peak concentration of NHC over the dosing interval. Plasma samples were collected at multiple time points pre-and post-administration and used to determine Cmax. Cmax of NHC was reported for participants receiving molnupiravir in Panels A and B.
Time Frame: Day -1: Predose and 12 hours postdose; Days 2, 5, and 6: 12 hours postdose; Days 4 and 7: predose and 0.5, 1.5, 4, 8, and 12 hours postdose
Population: All randomized participants in Panels A and B who received at least one dose of molnupiravir and received viral inoculation, with available measurements and without important protocol deviations. Per protocol, Panel C participants receiving placebo were not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel B: Molnupiravir Triggered Treatment
Number analyzed (Participants) | 38 | 36
ng/mL | 3640 (33.5) | 3010 (111.5)

31. Secondary Outcome: Panels A & B: Time to Maximum Plasma Concentration (Tmax) of NHC
Description: NHC is the pharmacologically active moiety of molnupiravir and therefore its primary pharmacokinetic measure. Tmax was defined as the time to peak concentration. Plasma samples were collected at multiple time points pre-and post-administration and used to determine Tmax. Tmax of NHC was reported for participants receiving molnupiravir in Panels A and B.
Time Frame: as for outcome 30
Population: as for outcome 30
Measure: Median (Full Range); unit: hr
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel B: Molnupiravir Triggered Treatment
Number analyzed (Participants) | 38 | 36
hr | 1.47 [1.33 to 1.97] | 1.48 [0.00 to 2.13]

32. Secondary Outcome: Panels A & B: Area Under the Plasma Concentration Curve From 0 to 12 Hours Postdose (AUC0-12) of NHC
Description: NHC is the pharmacologically active moiety of molnupiravir and therefore its primary pharmacokinetic measure. Plasma samples were collected at multiple time points pre-and post-administration and used to determine the area under the plasma concentration curve from time 0 to 12 hours (AUC0-12). AUC0-12 was reported for participants receiving molnupiravir in Panels A and B.
Time Frame: as for outcome 30
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel B: Molnupiravir Triggered Treatment
Number analyzed (Participants) | 38 | 36
hr*ng/mL | 9270 (28.4) | 8100 (87.9)

33. Secondary Outcome: Panels A & B: Trough Concentration (Ctrough) of NHC
Description: NHC is the pharmacologically active moiety of molnupiravir and therefore its primary pharmacokinetic measure. The trough concentration (Ctrough) was defined as the lowest concentration before the next dose. Plasma samples were collected at multiple time points pre-and post-administration and used to determine Cmax. Ctrough of NHC in plasma was reported for participants receiving molnupiravir in Panels A and B.
Time Frame: Day 2 at 12 hours predose (Panel A) or Day 6 at 12 hours predose (Panel B)
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel B: Molnupiravir Triggered Treatment
Number analyzed (Participants) | 38 | 36
ng/mL | 25.1 (55.6) | 19.8 (66.8)

ADVERSE EVENTS:
Time Frame: Day -1 up to Day 28
Description: All-Cause Mortality is reported for all randomized participants. Serious adverse events and non-serious (other) adverse events are reported for all participants that received at least one dose of study treatment.
Groups:
- Panel A: Molnupiravir Prophylaxis: Participants received molnupiravir 800 mg every 12 hours for 5 days beginning on Day -1, and were inoculated with RSV-A Memphis 37b on Day 0. Participants switched to placebo beginning on the evening of Day 4 to the morning of Day 10.
Arm/Group | Panel A: Molnupiravir Prophylaxis | Panel B: Molnupiravir Triggered Treatment | Panel C: Matched Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/36 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/36 | 0/40
Other Adverse Events (participants affected / at risk) | 1/39 | 2/36 | 0/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: Molnupiravir Prophylaxis (N=39) | Panel B: Molnupiravir Triggered Treatment (N=36) | Panel C: Matched Placebo (N=40)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Authorship will be determined by mutual agreement and in line with ICMJE authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT05559905/Prot_SAP_000.pdf